CLINICAL TRIAL: NCT04301154
Title: Phase I, Proof of Concept, Open-Label, Randomized Clinical Trial to Evaluate the Safety and Effects of Using Prime-boost HIVIS DNA and MVA-CMDR Vaccine Regimens With or Without Toll-like Receptor 4 Agonist on HIV Reservoirs in Perinatally HIV Infected Children and Youth
Brief Title: Safety and Effects of Using Prime-boost HIVIS DNA and MVA-CMDR Vaccine Regimens With or Without Toll-like Receptor 4 Agonist on HIV Reservoirs in Perinatally HIV Infected Children and Youth
Acronym: HVRRICANE
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Henry M. Jackson Foundation for the Advancement of Military Medicine (Other)
Collaborators: Bambino Gesù Hospital and Research Institute (Other); PENTA Foundation (Network); Johns Hopkins University (Other); University of Miami (Other); Leidos Biomedical Research, Inc. (Industry); Case Western Reserve University (Other); Karolinska Institutet (Other); Walter Reed Army Institute of Research (WRAIR) (U.S. Federal Agency); Armed Forces Research Institute of Medical Sciences, Thailand (Other Government); University of Padova (Other); Chulalongkorn University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RV534
Record Dates: First submitted 2020-03-02; First posted 2020-03-10 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-08

CONDITIONS: HIV Infections
Keywords: HIV reservoir; Perinatally HIV Infected Children; Vaccine
MeSH Terms: conditions — HIV Infections | interventions — human papillomavirus vaccine, L1 type 16, 18

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Arm 1 (n=10): HIVIS DNA / MVA-CMDR (Experimental): Arm 1 (n=10) will receive 1500 micrograms (0.5ml) HIVIS DNA IM by needle-free injection at weeks 0 and 4 followed by intramuscular (IM) needle injection of 1 X 108 IU/mL (1ml) MVA-CMDR at weeks 24 and 36 in the same arm as HIVIS DNA.
  Participants who have been randomized to receive HIVIS DNA and MVA-CMDR alone (ARM 1) will be administered Cervarix after week 72, the last study follow-up visit, if required.
  Interventions: Biological: HIVIS DNA/MVA-CMDR
- Arm 2 (n=10): HIVIS DNA + Cervarix/ / MVA-CMDR (Experimental): Arm 2 (n=10) will receive 0.5 ml of Cervarix IM by needle injection followed by 1500 micrograms (0.5ml) per injection of HIVIS DNA IM by a needle-free injection device in the skin above (proximal to) the Cervarix injection (within 1.5 cm). They will receive 1 X 108 IU/mL (1ml) MVA-CMDR IM by needle injection at weeks 24 and 36 in the same arm as HIVIS DNA. They will also receive 0.5 ml Cervarix at the time of the first MVACMDR injection in the opposite arm from the MVA injection at week 24.
  Interventions: Biological: HIVIS DNA + Cervarix and MVA-CMDR
- Arm 3 (n=5): Cervarix (Experimental): Arm 3 (n=5) will receive 0.5 ml of Cervarix by IM needle injection at weeks 0, 4 and 24.
  Interventions: Biological: Cervarix

INTERVENTIONS:
Biological: HIVIS DNA/MVA-CMDR — HIVIS DNA IM by needle-free injection at weeks 0 and 4 followed by intramuscular (IM) needle injection of 1 X 108 IU/mL (1ml) MVA-CMDR at weeks 24 and 36 in the same arm as HIVIS DNA.
  Arms: Arm 1 (n=10): HIVIS DNA / MVA-CMDR
Biological: HIVIS DNA + Cervarix and MVA-CMDR — Cervarix IM by needle injection followed by 1500 micrograms (0.5ml) per injection of HIVIS DNA IM by a needle-free injection device in the skin above (proximal to) the Cervarix injection (within 1.5 cm). They will receive 1 X 108 IU/mL (1ml) MVA-CMDR IM by needle injection at weeks 24 and 36 in the same arm as HIVIS DNA. They will also receive 0.5 ml Cervarix at the time of the first MVACMDR injection in the opposite arm from the MVA injection at week 24.
  Arms: Arm 2 (n=10): HIVIS DNA + Cervarix/ / MVA-CMDR
Biological: Cervarix — Cervarix by IM needle injection at weeks 0, 4 and 24.
  Arms: Arm 3 (n=5): Cervarix

SUMMARY:
Phase I, Proof of Concept, Open-Label, Randomized Clinical Trial to Evaluate the Safety and Effects of Using Prime-boost HIVIS DNA and MVA-CMDR Vaccine Regimens with or without Toll-like Receptor 4 Agonist on HIV Reservoirs in Perinatally HIV Infected Children and Youth

DETAILED DESCRIPTION:
HIVIS DNA and MVA-CMDR vaccines induce immune responses important for clearing infected cells: broad HIV-specific CD8+ cytotoxic T cells, potent antibodydependent cellular cytotoxicity (ADCC), and binding antibody (Ab) and neutralizing antibody (NAb). The study include early treated children because of their healthy immunity and small HIV reservoirs. Giving licensed vaccine, Cervarix®, against human papilloma virus (HPV) that contains toll-like receptor (TLR) 4 agonist with HIVIS DNA could increase DNA antigen loading on dendritic cells and promote adaptive immune responses to the HIV vaccine.

ELIGIBILITY:
Inclusion criteria:

1. HIV perinatally infected
2. Know their HIV+ status
3. Initiated ART prior to 6 months of age
4. Male and female ≥ 9 years old
5. In generally good health
6. Plasma viral load < 200 copies/ml on ART at screening
7. CD4 count above 400 cells/mm3 at screening
8. Participants of childbearing potential who are sexually active must be willing to practice effective contraception during the study
9. Negative urine β-HCG (human chorionic gonadotropin) pregnancy test for any female of childbearing age (post-menarche)
10. Availability for follow-up for planned duration of the study
11. Passing a test of understanding is required for participants ≥ 18 years old or the parent(s)/legal representative of participants < 18 years old before consent.
12. Written informed consent from participants ≥ 18 years old or parent(s)/legal representative of participants < 18 years old. Assent by participants aged 9-17 years old will also be required.
13. Laboratory criteria within 8 weeks prior to enrollment

    * Hb >11.0 g/dl
    * White blood cell count >3000 cells/mm3
    * Platelets >125,000/ mm3
    * ALT <1.5 x upper limit of normal
    * Creatinine <1.5 x upper limit of normal

Exclusion criteria:

1. Participants who experienced virological failure necessitating ART modifications
2. Participants who had ART interruption that lasted >2 weeks
3. Prior or current pancreatitis or history of alcohol abuse.
4. Systemic cortisone treatment within the past 30 days
5. Participants coinfected with chronic hepatitis B (Hepatitis B surface antigen, HBsAg+) or hepatitis C (Hepatitis C antibody, HCV Ab+) at screening
6. Participants with signs of autoimmune diseases
7. Participants with history of myocarditis
8. Participants on any immune modulating or investigational drug
9. Pregnant or breastfeeding female

Min Age: 9 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2022-02-18 (Actual); Primary Completion 2023-10-16 (Actual); Study Completion 2023-10-16 (Actual)

PRIMARY OUTCOMES:
Solicited and unsolicited serious adverse events | through study completion, an average of 1 year
  Safety
Frequencies of CD4+ T cells that produce Tat/Rev transcription (tat/rev RNA+ cells/106 CD4+ T cells) | Change from Baseline at week 24, 36, 48, 60, 72
  Efficacy
HIV DNA (copies/106 CD4+ T cells) | Change from Baseline at week 28, 48
  Efficacy

SECONDARY OUTCOMES:
Solicited and unsolicited non-serious adverse events | through study completion, an average of 1 year
  Safety
Unspliced and multiply-spliced RNA+ cells/1000 ng cellular RNA | Week 24, 36, 48, 60, 72
  Efficacy
IUPM from total CD4+ T cells in blood by QVOA | Week 24, 36, 48, 60, 72
  Efficacy
Plasma HIV RNA by SCA | Week 24, 36, 48, 60, 72
  Efficacy
HIV-specific CD8+ and CD4+ T cells | Week 28, 48
  Immunogicity
ADCC | Week 28, 48
  Immunogicity
Binding and neutralizing Ab | Week 28, 48
  Immunogicity
Global gene expression on PBMCs by RNA seq | Week 28, 48
  immune response
Gene expression on HIV-specific CD8+ and CD4+ T cells | Week 28, 48
  immune response

CONTACTS AND LOCATIONS:
Overall Officials: Merlin Robb, MD, Study Chair — Henry M. Jackson Foundation for the Advancement of Military Medicine
Locations (1):
- Stellenbosch University, Tygerberg Hills, Cape Town, South Africa

IPD SHARING:
Plan to Share IPD: No